CLINICAL TRIAL: NCT01530919
Title: Minimally Invasive Radioguided Parathyroidectomy
Acronym: MIRP
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: Norton Healthcare (Other); Jewish Hospital and St. Mary's Healthcare (Other)
Responsible Party: Principal Investigator, Michael B. Flynn, MD, Professor, University of Louisville
Other Study IDs: 291.97
Record Dates: First submitted 2011-11-30; First posted 2012-02-10 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Small portion of abnormal parathyroid gland that is removed during surgery is frozen and stored for future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parathyroid surgery: Database of patients who have undergone minimally invasive radioguided parathyroidectomy
  Interventions: Procedure: Minimally invasive radioguided parathyroidectomy

INTERVENTIONS:
Procedure: Minimally invasive radioguided parathyroidectomy — After the patient is prepared for surgery and under local anesthesia, the initial incision by the surgeon will be 2-3 cm. The surgeon will dissect in the designated quadrant until the parathyroid gland is identified.

SUMMARY:
The main purpose of this research study is to evaluate the effectiveness of a minimally invasive surgical approach to removing parathyroid gland(s). The researchers are also interested in analyzing abnormal parathyroid tissue for changes in genes and proteins that may contribute to overactive parathyroid gland(s).

DETAILED DESCRIPTION:
The specific aims of this study are to determine the safety and efficacy of minimally invasive radioguided parathyroidectomy, to determine the positive and negative predictive value of sestamibi scanning to detect parathyroid adenomas, and to differentiate adenomas from parathyroid hyperplasia. In addition, this study aims to determine the value of intraoperative parathyroid hormone assay to verify biochemical cure of primary hyperparathyroidism, to determine whether minimally invasive radioguided parathyroidectomy is cos-effective, and to collect abnormal parathyroid tissue at the time of surgery for tissue analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with biochemical evidence of primary hyperparathyroidism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and minors diagnosed with primary hyperparathyroidism that will be having minimally invasive radioguided parathyroidectomy surgery to correct this condition at either Norton Hospital, University of Louisville Hospital or Jewish Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 856 (Actual)
Dates: Start 1998-09; Primary Completion 2009-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The positive and negative predictive value of sestamibi scanning to detect parathyroid adenomas. | 2-3days

SECONDARY OUTCOMES:
The value of intraoperative parathyroid hormone assay to verify biochemical cure or primary hyperparathyroidism | 2-3 days
Collection of abnormal parathyroid tissue at the time of surgery for tissue analysis | day of surgery (1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Flynn, M.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Result] Quillo AR, Bumpous JM, Goldstein RE, Fleming MM, Flynn MB. Minimally invasive parathyroid surgery, the Norman 20% rule: is it valid? Am Surg. 2011 Apr;77(4):484-7. PMID 21679561
- [Result] Grady JA, Bumpous JM, Fleming MM, Flynn MB, Turbiner E, Lentsch EJ, Ziegler CH. Advantages of a targeted approach in minimally invasive radioguided parathyroidectomy surgery for primary hyperparathyroidism. Laryngoscope. 2006 Mar;116(3):431-5. doi: 10.1097/01.mlg.0000195288.06601.18. PMID 16540904
- [Result] Flynn MB, Quayyum M, Goldstein RE, Bumpous JM. Outpatient parathyroid surgery: ten-year experience: is it safe? Am Surg. 2015 May;81(5):472-7. PMID 25975331
- [Result] Flynn MB, Bumpous JM, Schill K, McMasters KM. Minimally invasive radioguided parathyroidectomy. J Am Coll Surg. 2000 Jul;191(1):24-31. doi: 10.1016/s1072-7515(00)00297-0. PMID 10898180
- [Result] Hutchinson JR, Yandell DW, Bumpous JM, Fleming MM, Flynn MB. Three-year financial analysis of minimally invasive radio-guided parathyroidectomy. Am Surg. 2004 Dec;70(12):1112-5. PMID 15663056
- [Result] Goldstein RE, Carter WM 2nd, Fleming M, Bumpous J, Lentsch E, Rice M, Flynn M. Unilateral cervical surgical exploration aided by intraoperative parathyroid hormone monitoring in patients with primary hyperparathyroidism and equivocal sestamibi scan results. Arch Surg. 2006 Jun;141(6):552-7; discussion 557-9. doi: 10.1001/archsurg.141.6.552. PMID 16785355
- [Result] Kartha SS, Chacko CE, Bumpous JM, Fleming M, Lentsch EJ, Flynn MB. Toxic metabolic encephalopathy after parathyroidectomy with methylene blue localization. Otolaryngol Head Neck Surg. 2006 Nov;135(5):765-8. doi: 10.1016/j.otohns.2006.05.026. PMID 17071309
- [Result] Conn CA, Clark J, Bumpous J, Goldstein R, Fleming M, Flynn MB. Hypocalcemia after neck exploration for untreated primary hyperparathyroidism. Am Surg. 2006 Dec;72(12):1234-7. PMID 17216827
- [Result] Han N, Bumpous JM, Goldstein RE, Fleming MM, Flynn MB. Intra-operative parathyroid identification using methylene blue in parathyroid surgery. Am Surg. 2007 Aug;73(8):820-3. PMID 17879694
- [Result] Stephen ET, Quillo AR, Lewis KE, Harden FL, Bumpous JM, Flynn MB, Callender GG. Operative failure rate and documentation of family history in young patients undergoing focused parathyroidectomy for primary hyperparathyroidism. Am Surg. 2015 Jun;81(6):585-90. PMID 26031271
- [Result] Bumpous JM, Goldstein RL, Flynn MB. Surgical and calcium outcomes in 427 patients treated prospectively in an image-guided and intraoperative PTH (IOPTH) supplemented protocol for primary hyperparathyroidism: outcomes and opportunities. Laryngoscope. 2009 Feb;119(2):300-6. doi: 10.1002/lary.20049. PMID 19160424
- [Result] Young VN, Osborne KM, Fleming MM, Flynn MB, Goldstein RE, Bumpous JM. Parathyroidectomy in the elderly population: does age really matter? Laryngoscope. 2010 Feb;120(2):247-52. doi: 10.1002/lary.20706. PMID 19950385